CLINICAL TRIAL: NCT02008422
Title: A Randomized, Open and Control Clinical Study of Endostar Injection Concomitant With SOX Protocols in Treating Advanced Gastric Cancer
Brief Title: Clinical Study of Endostar Injection Concomitant With SOX Protocols to Treat Advanced Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tang Xushan (Other)
Responsible Party: Sponsor-Investigator, Tang Xushan, Xinjiang Medical University, Xinjiang Medical University
Organization: Xinjiang Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XinjiangMU (006)
Record Dates: First submitted 2013-11-27; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; gimeracil; potassium oxonate; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxaliplatin & Endostar injection (Experimental): Oxaliplatin, 130 mg/m2 , iv, 3-4h, d1; Gimeracil and Oteracil Potassium Capsules, 40 mg/m2, po., Bid., d1-14; Endostar injection, 7.5 mg/m2/d, 2 mL/h continuous pumping into vein, d1-10; 21 d as a cycle.
  Interventions: Drug: Oxaliplatin; Drug: Gimeracil and Oteracil Potassium Capsule; Drug: Endostar injection
- Oxaliplatin (Active Comparator): Oxaliplatin, 130 mg/m2 , iv, 3-4h, d1; Gimeracil and Oteracil Potassium Capsules, 40 mg/m2, po., Bid., d1-14, 21 d as a cycle.
  Interventions: Drug: Oxaliplatin; Drug: Gimeracil and Oteracil Potassium Capsule

INTERVENTIONS:
Drug: Oxaliplatin — 130mg/m2 , iv, 3-4h, d1, 21 d as a cycle.
  Other Names: L-OHP
Drug: Gimeracil and Oteracil Potassium Capsule — 40 mg/m2, po., Bid., d1-14, 21 d as a cycle.
  Other Names: Tegafur Gimeracil Oteracil Potassium Capsule
Drug: Endostar injection — 7.5 mg/m2/d, 2 mL/h continuous pumping into vein, d1-10, 21 d as a cycle.
  Other Names: rh-Endostatin
  Arms: Oxaliplatin & Endostar injection

SUMMARY:
The primary objectives of this control, single-center clinical study of EndostarTM Injection with/without SOX protocols to treat advanced gastric cancer were to evaluate the clinical response rate of Endostar injection concomitant with SOX on patients with advanced gastric cancer, observe the progression-free survival time (PFS) of tumor and evaluate the safety and tolerance of Endostar injection, while the secondary objectives were to observe the influence of Endostar injection on chemotherapy-induced adverse reactions and evaluate the overall survival time of EndostarTM injection concomitant with SOX on patients with advanced gastric cancer by evaluating the response rate (RR) clinical benefit rate (CBR), progression-free survival (PFS) and overall survival (OS).

DETAILED DESCRIPTION:
Multiple pre-clinical studies have indicated that in dozens of animal tumor models and human tumor-metastatic mice tumor models, the effective rate of Endostar was 47%～91% in daily dosage of 10～100mg/kg, and covered human commonly seen malignant tumors, such as lung cancer, gastric cancer, breast cancer, colorectal cancer, hepatic cancer, malignant melanoma and non-Hodgkin's lymphoma, etc.. The development and progression of gastric cancer was in association with angiogenesis. An animal research observed the influence of Endostar on tumor strains in nude mice with gastric cancer, and the results showed that tumor size shrunk rapidly and the expressions of VEGF, bFGF, VEGF-C, VEGFR-3, bcl-2 and PDGF decreased significantly after treatment in experimental group, demonstrating that Endostar could reduce angiogenesis, increase tumor cell apoptosis and inhibit tumor growth in gastric cancer. An investigation of small-sample Endostar concomitant with chemotherapy on patients with advanced gastric cancer primarily indicated the efficacy and feasibility of Endostar concomitant with chemotherapy in treating gastric cancer.

With the expanded application of Endostar in clinic, it also obtains certain effect in treating patients with lung cancer and colorectal cancer. The safety, efficacy, evaluation of relationship between benefit and risk in common or special population as well as the modified dosage of administration of Endostar in wide application should be further explored to provide sufficient scientifical basis for the safety, efficacy, applicable rule in special population and investigation of optimal administrative protocols for Endostar in wide application.

This control, single-center clinical study of EndostarTM Injection with/without SOX protocols to treat advanced gastric cancer was conducted to explore the feasibility, efficacy and safety of Endostar concomitant with SOX protocols, and to provide more evidence-based medical basis for the clinical application of Endostar.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18～70 years;
* Performance status (PS) of Eastern Cooperative Oncology Group (ECOG) was 0～1 or KPS scores were 60-100 scores;
* Patients who were diagnosed with recurrent and metastatic advanced gastric cancer by histopathology and CT;
* Patients who had more than 1 measurable nidus (common CT or MRI scanning ≥20 mm, spiral CT scanning ≥10 mm);
* Patients who had no severe dysfunction of important organs, and were normal in blood routine test, hepatorenal function, electrolytes and cardiac function, with white blood cell count≥4.0×109/L, neutrophil count≥1.5×109/L, platelet count≥100×109/L, hemoglobin≥95g/L, serum bilirubin≤1.5 folds of upper normal limit, Alanine transaminase and glutamic oxalacetic transaminase ≤2 folds of upper normal limit, and serum creatinine≤1.5mg/dl.
* Estimated survival time was above 3 months;
* Patients who were well acknowledged of this study and signed the informed consent forms.

Exclusion Criteria:

* Patients who received whole body treatment of metastatic gastric cancer previously;
* Patients who underwent surgeries within 4 weeks before this study;
* Patients who had allergic constitutions or were allergic to biological products of proteins and to any medicine used in this study;
* Female patients in gestation or lactation period, or those who were interfile but received no contraception measures;
* Patients who were with other symptoms unsuitable to this study;
* Patients who were treated by other anti-tumor methods at that time;
* Patients who had no measurable nidus;
* Patients who had one of the following conditions: uncontrolled metastatic nidus in central nervous system, dysfunction of important organs, severe cardiac diseases (including congestive heart failure, uncontrollable arrhythmia, angina pectoris needed long-term drug treatment, valvular heart diseases and myocardial infarction), hypertension, women in gestation or lactation period, protracted infectious wound as well as uncontrollable psychosis history.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Response rate (RR) | The patients were followed up for 3 years.
  * Clinical RR=(CR＋PR)/total cases×100%;
  * Complete remission (CR): all visible nidi disappeared;
  * Partial remission (PR): the decreased total length of diameter of baseline nidus≥30%;
clinical benefit rate (CBR) | The patients were followed up for 3 years.
  * Clinical CBR＝(CR＋PR＋SD)/total cases×100%
  * Complete remission (CR): all visible nidi disappeared;
  * Stable disease (SD): the total length of diameter of baseline nidus decreased<that in PR or increased <that in PD.-Progressive disease (PD): the increased total length of diameter of baseline nidus≥30% or new nidus was presented;
progression-free survival (PFS) | The patients were followed up for 3 years
  PFS was from randomization to tumor progression or death.

SECONDARY OUTCOMES:
overall survival (OS) | The patients were followed up for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tang Yong, Professor, Study Director — Cnacer Hospital of Xinjiang Medical University
Locations (1):
- Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China